CLINICAL TRIAL: NCT01405508
Title: A Multi-center, Open-label, Four-arm, Randomized Trial Evaluating the Safety and Tolerability of Brivaracetam Intravenous Infusion and Bolus, Administered in BID Regimen as an Adjunctive Antiepileptic Treatment in Subjects From 16 to 70 Years Suffering From Epilepsy
Brief Title: Safety and Tolerability of Intravenous Brivaracetam (Infusion or Bolus) as Adjunctive Antiepileptic Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N01258; 2008-004714-27 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2016-07

CONDITIONS: Epilepsy
Keywords: N01258; Brivaracetam; Epilepsy; IV; intravenous
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo tablets / Brivaracetam bolus (Experimental): Subjects will receive Placebo (PBO) tablets for one week followed by Brivaracetam (BRV) bolus for 4.5 days.
  Down-Titration:
  * If subject discontinues the study during the Run-In Period, then the subject will receive the treatment that he/she was assigned during Run-In
  * If subject discontinues during the Evaluation Period or after Day 12, the subject will receive Placebo tablets during Down-Titration:
  Tablets will be provided for 4 weeks; 75 mg / intake BID for the first week, 50 mg / intake BID for the second week, 25 mg / intake BID for the third week, 10 mg / intake BID for the fourth week
  Interventions: Drug: Brivaracetam bolus; Other: Placebo
- Brivaracetam (BRV) tablets / BRV bolus (Experimental): Subjects will receive Brivaracetam (BRV) tablets for one week followed by BRV bolus for 4.5 days.
  Down-Titration:
  * If subject discontinues the study during the Run-In Period, then the subject will receive the treatment that he/she was assigned during Run-In
  * If subject discontinues during the Evaluation Period or after Day 12, the subject will receive BRV tablets during Down-Titration:
  Tablets will be provided for 4 weeks; 75 mg / intake BID for the first week, 50 mg / intake BID for the second week, 25 mg / intake BID for the third week, 10 mg / intake bid for the fourth week
  Interventions: Drug: Brivaracetam tablets; Drug: Brivaracetam bolus
- Placebo tablets / Brivaracetam infusion (Experimental): Subjects will receive Placebo (PBO) tablets for one week followed by Brivaracetam (BRV) intravenous infusion for 4.5 days.
  Down-Titration:
  * If subject discontinues the study during the Run-In Period, then the subject will receive the treatment that he/she was assigned during Run-In
  * If subject discontinues during the Evaluation Period or after Day 12, the subject will receive BRV tablets during Down-Titration:
  Tablets will be provided for 4 weeks; 75 mg / intake BID for the first week, 50 mg / intake BID for the second week, 25 mg / intake BID for the third week, 10 mg / intake BID for the fourth week
  Interventions: Drug: Brivaracetam infusion; Other: Placebo
- Brivaracetam (BRV) tablets / BRV infusion (Experimental): Subjects will receive Brivaracetam (BRV) tablets for one week followed by Brivaracetam intravenous infusion for 4.5 days.
  Down-Titration:
  * If subject discontinues the study during the Run-In Period, then the subject will receive the treatment that he/she was assigned during Run-In
  * If subject discontinues during the Evaluation Period or after Day 12, the subject will receive BRV tablets during Down-Titration:
  Tablets will be provided for 4 weeks; 75 mg / intake BID for the first week, 50 mg / intake BID for the second week, 25 mg / intake BID for the third week, 10 mg / intake BID for the fourth week
  Interventions: Drug: Brivaracetam tablets; Drug: Brivaracetam infusion

INTERVENTIONS:
Drug: Brivaracetam tablets — 100 mg, intake twice daily (BID) for 7 days during Run-In Period
  Arms: Brivaracetam (BRV) tablets / BRV bolus; Brivaracetam (BRV) tablets / BRV infusion
Drug: Brivaracetam bolus — 10 mL (= 100 mg) of Brivaracetam administered intravenously over 2 minutes twice daily (BID) during Evaluation Period
  Arms: Brivaracetam (BRV) tablets / BRV bolus; Placebo tablets / Brivaracetam bolus
Drug: Brivaracetam infusion — 10 mL (= 100 mg) of Brivaracetam diluted in 90 mL 0.9 % isotonic saline sterile solution for intravenous administration infused over 15 minutes twice daily (BID) during Evaluation Period
  Arms: Brivaracetam (BRV) tablets / BRV infusion; Placebo tablets / Brivaracetam infusion
Other: Placebo — 100 mg twice daily (BID) for 7 days during Run-In Period
  Arms: Placebo tablets / Brivaracetam bolus; Placebo tablets / Brivaracetam infusion

SUMMARY:
This is a multicenter, open-label, 4-arm, randomized, parallel-group study to evaluate safety and tolerability of Brivaracetam Intravenous (BRV iv) as adjunctive treatment for adults with epilepsy according to an initiation or a conversion scheme, during repeated dosing (100 mg/administration twice daily for 4.5 days).

DETAILED DESCRIPTION:
Eligible subjects will be randomized in a 1:1:1:1 ratio to the 4 treatment arms

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board/Independent Ethics Committee (IRB/IEC) approved written Informed Consent form signed and dated by the subject or by parent(s) or legal representative
* Subjects from 16 to 70 years
* Subjects with a body weight of >/= 40 kg
* Female subjects without childbearing potential or female subjects with childbearing potential if they use a medically accepted contraceptive method
* Subject/legal representative considered as reliable and capable of adhering to the protocol
* Subjects with well-characterized focal or generalized epilepsy or epileptic syndrome
* Subjects with a history of partial-onset seizures whether or not secondarily generalized or primary generalized seizures
* Subjects being uncontrolled while treated with 1 to 2 permitted concomitant antiepileptic drugs (AEDs)
* Permitted concomitant antiepileptic drugs (AEDs) and vagus nerve stimulation (VNS) being stable and at optimal dosage for the subject from at least 1 month before Visit 1 and expected to be kept stable during the Run-In and Evaluation Periods

Exclusion Criteria:

* Mentally impaired subjects unable to understand the study purpose
* History or presence of status epilepticus during 1 year preceding Visit 1 or Baseline
* Subjects on felbamate with less than 18 months continuous exposure before Visit 1
* Subjects currently on vigabatrin
* Subject taking any drug with possible relevant central nervous system effects except is stable from at least 1 month before Visit 1 and expected to be kept stable during the trial
* Subjects taking any drug that may significantly influence the metabolism of Brivaracetam (BRV) except if the dose has been kept stable at least 1 month before Visit 1, and is expected to be kept stable during the trial
* History of cerebrovascular accident in the last 6 months
* Subjects suffering from severe cardiovascular disease or peripheral vascular disease
* Presence of any sign suggesting rapidly progressing brain disorder or brain tumor
* Any clinical conditions which impair reliable participation in the study or necessitate the use of medication not allowed by protocol
* Presence of a terminal illness
* Presence of a serious infection
* Subjects with a history of sever adverse hematologic reaction to any drug
* Subjects suffering from severe disturbance of hemostasis
* Impaired hepatic function: alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyltransferase (GGT) values of more than 3 times the upper limit of the reference range
* Subjects having clinically significant deviations from reference range values for laboratory parameters: creatinine clearance calculated < 50 ml / min, platelets < 100,000 / µL, or neutrophil cells < 1,800 / µL
* Clinically significant electrocardiogram (ECG) abnormalities according to the Investigator
* History of suicide attempt
* In the Investigator's medical judgment, any current suicidal ideation or other serious psychiatric disorders requiring of having required hospitalization or medication
* Known allergic reaction or intolerance to pyrrolidone derivatives and / or investigational product excipients
* Known multiple drug allergies or severe drug allergy
* Pregnant or lactating women
* Known alcohol or drug addiction or abuse within the last 2 years
* Subject institutionalized under judicial decision
* Problems of venous accessibility
* Subject taking part in another clinical / pharmacological study in the month preceding enrollment (Visit 1)
* Investigators, coinvestigators, their spouses or children, or any study collaborators
* Subjects previously treated with Brivaracetam (BRV)
* Subject previously screened within this study

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (17):
- United States (8):
  - 001, Phoenix, Arizona
  - 775, Little Rock, Arkansas
  - 780, Lexington, Kentucky
  - 008, Bethesda, Maryland
  - 778, Columbus, Ohio
  - 776, Nashville, Tennessee
  - 777, Dallas, Texas
  - 036, Charlottesville, Virginia
- Czechia (4):
  - 917, Brno
  - 915, Hradec Králové
  - 916, Kroměříž
  - 913, Ostrava Poruba
- Germany (2):
  - 332, Bielefeld
  - 903, Bonn
- Poland (3):
  - 795, Katowice
  - 479, Poznan
  - 794, Warsaw

REFERENCES:
- [Derived] Toledo M, Brandt C, Quarato PP, Schulz AL, Cleveland JM, Wagener G, Klein P. Long-term safety, efficacy, and quality of life during adjunctive brivaracetam treatment in patients with uncontrolled epilepsy: An open-label follow-up trial. Epilepsy Behav. 2021 May;118:107897. doi: 10.1016/j.yebeh.2021.107897. Epub 2021 Mar 27. PMID 33780735

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to recruit patients in August 2011 and concluded in July 2012.
  105 subjects were randomized to 4 different treatment groups.
Pre-assignment Details: Participant Flow refers to the Randomized Set (RS).
Period: Overall Study
Arm/Group | Placebo Tablets / Brivaracetam Bolus | Placebo Tablets / Brivaracetam Infusion | Brivaracetam (BRV) Tablets / BRV Bolus | Brivaracetam (BRV) Tablets / BRV Infusion
Started | 26 | 26 | 27 | 26
Completed | 25 | 25 | 27 | 26
Not Completed | 1 | 1 | 0 | 0
Not completed — AE, non-serious non-fatal | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characetristics refer to the Safety Population consisting of all subjects who took at least 1 dose of study drug.
Arm/Group | Placebo Tablets / Brivaracetam Bolus | Placebo Tablets / Brivaracetam Infusion | Brivaracetam (BRV) Tablets / BRV Bolus | Brivaracetam (BRV) Tablets / BRV Infusion | Total Title
Number analyzed (Participants) | 26 | 26 | 27 | 26 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 25 | 27 | 25 | 103
  >=65 years | 0 | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (12.2) | 39.5 (14.4) | 42.0 (9.2) | 44.4 (12.6) | 41.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 17 | 17 | 56
  Male | 14 | 16 | 10 | 9 | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Treatment-emergent Adverse Event During the Study (Maximum 40 Days)
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: 40 days
Population: Safety Population consisting of all subjects who took at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo Tablets / Brivaracetam Bolus | Placebo Tablets / Brivaracetam Infusion | Brivaracetam (BRV) Tablets / BRV Bolus | Brivaracetam (BRV) Tablets / BRV Infusion
Number analyzed (Participants) | 26 | 26 | 27 | 26
Participants | 20 | 19 | 21 | 20

2. Secondary Outcome: Number of Subjects Who Withdrew Due to a Treatment-emergent Adverse Event During the Study (Maximum 40 Days)
Description: as for outcome 1
Time Frame: 40 days
Population: Safety Population consisting of all subjects who took at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo Tablets / Brivaracetam Bolus | Placebo Tablets / Brivaracetam Infusion | Brivaracetam (BRV) Tablets / BRV Bolus | Brivaracetam (BRV) Tablets / BRV Infusion
Number analyzed (Participants) | 26 | 26 | 27 | 26
Participants | 1 | 1 | 0 | 0

3. Secondary Outcome: Number of Subjects With at Least One Injection-related Treatment-emergent Adverse Event (TEAE) During the Evaluation Period.
Description: as for outcome 1
Time Frame: 4.5-day Evaluation Period
Population: Safety Population consisting of all subjects who took at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo Tablets / Brivaracetam Bolus | Placebo Tablets / Brivaracetam Infusion | Brivaracetam (BRV) Tablets / BRV Bolus | Brivaracetam (BRV) Tablets / BRV Infusion
Number analyzed (Participants) | 26 | 26 | 27 | 26
Participants | 1 | 3 | 4 | 3

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Baseline over Run-In (Day 1) and Evaluation Period (Day 8 to Day 12) to the Safety Visit or Early Discontinuation Visit (up to 54 days).
Description: Adverse Events refer to the Safety Population consisting of all subjects who took at least 1 dose of study drug.
Arm/Group | Placebo Tablets / Brivaracetam Bolus | Placebo Tablets / Brivaracetam Infusion | Brivaracetam (BRV) Tablets / BRV Bolus | Brivaracetam (BRV) Tablets / BRV Infusion
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 17/26 | 15/26 | 15/27 | 14/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Tablets / Brivaracetam Bolus (N=26) | Placebo Tablets / Brivaracetam Infusion (N=26) | Brivaracetam (BRV) Tablets / BRV Bolus (N=27) | Brivaracetam (BRV) Tablets / BRV Infusion (N=26)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (4) | 3 (4) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 8 (8) | 7 (7) | 7 (9) | 9 (10)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days